CLINICAL TRIAL: NCT02708225
Title: The Influence of Medical Clowns on the Performance of Pulmonary Function Tests Among Preschooler Children
Acronym: clowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0026-15
Record Dates: First submitted 2015-09-29; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Asthma; Pneumonia
MeSH Terms: conditions — Asthma; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- interventional - with a medical clown (Experimental): will perform pulmonary function test without the presence of a clown and an hour later will re-do the test with a medical clown present
  Interventions: Behavioral: medical clown
- non interventional (No Intervention): will perform pulmonary function test without the presence of a clown and an hour later will re-do the test without a medical clown present

INTERVENTIONS:
Behavioral: medical clown — a medical clown will assist the child during the performance of pulmonary function test
  Arms: interventional - with a medical clown

SUMMARY:
Medical clowns are known to assist in relaxing children and allowing better cooperation during performance of medical procedures.

The ability of medical clowns to improve the motivation of children to perform active tasks was never examined to date.

The investigators would like to examine the influence of the clowns' presence on the performance of pulmonary function test.

DETAILED DESCRIPTION:
The investigators would like to evaluate the performance of pulmonary function tests among preschool children aged 3-6 years.

Overall 200 children will participate.

The children will perform pulmonary function test without a clown present.

About an hour later half of them will perform the exam again with a medical clown assistance and the second half will repeat the examination without a clown present the differences between the performance will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* children visiting the pediatric pulmonology clinic
* parents signed informed consent

Exclusion Criteria:

* medical or neurological diseases not allowing performance of pulmonary function tests
* parents refusal

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
length of experium (seconds) | through study completion; estimate 1 year
  length of experium (seconds)
FEV1 (%predicted) | through study completion; estimate 1 year
  forced experiom volume within 1 second (% predicted)

CONTACTS AND LOCATIONS:
Overall Officials: vers NIR, MD, Principal Investigator — Hillel Yaffe Medical Center

IPD SHARING:
Plan to Share IPD: Yes
study results and conclusions will be published